CLINICAL TRIAL: NCT03607747
Title: Longitudinal Change of Arterial Stiffness Indices in Relation to Ambulatory Aortic and Branchial Pressure in Long Term Peritoneal Dialysis Patients
Brief Title: Relationship Between Blood Pressure and Pulse Wave Velocity Measurements in Peritoneal Dialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Vaios Vasileios, Principal Investigator, Division of Nephrology and Hypertension, 1st Department of Medicine, AHEPA University Hospital, Aristotle University Of Thessaloniki
Other Study IDs: MedAuth
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: End Stage Renal Disease; Peritoneal Dialysis; Arterial Sclerosis
Keywords: Arterial Stiffness; Pulse Wave Velocity; Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the relationship between Ambulatory Aortic and Branchial blood pressure vs Office blood pressure measurements with the changes in arterial stiffness indices, in long-term Peritoneal Dialysis (PD) patients. These parameters will be monitored both cross-sectionally at the start of the study and prospectively over a 6 month period.

DETAILED DESCRIPTION:
All participants will be monitored over a 6 month period during which 7 monthly visits will be performed. Brachial and aortic blood pressure (BP), wave reflection and arterial stiffness indices will be assessed with the brachial cuff-based oscillometric device Mobil-O-Graph NG (IEM, Stolberg, Germany). The above hemodynamic and arterial wall parameters will be measured for 24-hours on visits 1 (baseline) and 7 (month 6). The monitor will be set to obtain recordings 3 times/hour from 11:00 pm to 06:59 am and 2 times/hour from 07:00 am to 10:59 pm. Measurements will be used for the analysis if >80% of recordings were valid with no more than two non-consecutive day hours with fewer than two valid measurements, and no more than one night hour without valid recording, according to recommendations for ambulatory BP monitoring. Bioelectrical Impendance Analysis (BIA) with the Fresenius Body Composition Monitor (BCM - Fresenius Medical Care, Bad Homberg, Germany) will be performed on visits 1, 4 and 6 in order to assess the hydration status and body composition parameters of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or higher
2. Renal replacement therapy with Peritoneal Dialysis (Automated or Continuous Ambulatory) for at least 3 months prior to study enrollment
3. Patient to have provided informed written consent

Exclusion Criteria:

1. Ongoing atrial fibrillation
2. Hospitalization for acute myocardial infarction, unstable angina or acute ischemic stroke within the 3 previous months
3. Recent episode of PD-related peritonitis or exit site infection 1 month or less prior to study enrollment
4. Bilateral functioning or non-functioning arteriovenous fistula (AVF) and/or arteriovenous graft (AVG) used earlier for dialysis access in patients previously treated with hemodialysis
5. Body mass index (BMI) of >40 kg/m2
6. History of malignancy or any other clinical condition associated with very poor prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients with end stage renal disease receiving peritoneal dialysis for more than 3 months.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
24-hour ambulatory Branchial vs office Branchial Systolic BP (SBP) as determinants of Pulse Wave Velocity | 6 months
  24-hour ambulatory Branchial vs office Branchial SBP: which measurement correlates stronger with the changes in Pulse Wave Velocity over a 6 month period

SECONDARY OUTCOMES:
24-hour ambulatory Aortic SBP vs 24-hour ambulatory Branchial SBP as determinants of Pulse Wave Velocity | 6 months
  24-hour ambulatory Aortic SBP vs 24-hour ambulatory Branchial SBP: which measurement correlates stronger with the changes in Pulse Wave Velocity over a 6 month period
Short-term variability of 24-hour ambulatory Branchial and Aortic SBP as a determinant of Pulse Wave Velocity | 0, 6 months
  Assessing the correlation between the short-term variability of 24-hour ambulatory Branchial and Aortic SBP with the changes in Pulse Wave Velocity at the start of the study and over a 6 month period
Visit-to-visit variability of Branchial SBP as a determinant of Pulse Wave Velocity | 6 months
  Assessing the predictive value of visit-to-visit variability of Branchial SBP for the changes in Pulse Wave Velocity over a 6 month period
Office blood pressure monitoring for the diagnosis of hypertension in peritoneal dialysis patients | 0, 6 months
  Assessing whether or not office blood pressure measurements can diagnose hypertension or control of hypertension, based on the 24-hour ambulatory recordings
The effect of overhydration on 24-hour ambulatory measurements | 0, 3, 6 months
  The correlation between overhydration (defined by the measurement of fluid status using Bioelectrical Impendence Analysis) and the 24-hour ambulatory Aortic and Branchial SBP measurements at the start of the study and over a 6 month period

CONTACTS AND LOCATIONS:
Overall Officials: Vassilios Liakopoulos, MD, PhD, Study Director — Department of Medicine, Aristotle University of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Tonelli M, Wiebe N, Culleton B, House A, Rabbat C, Fok M, McAlister F, Garg AX. Chronic kidney disease and mortality risk: a systematic review. J Am Soc Nephrol. 2006 Jul;17(7):2034-47. doi: 10.1681/ASN.2005101085. Epub 2006 May 31. PMID 16738019
- [Background] Briet M, Boutouyrie P, Laurent S, London GM. Arterial stiffness and pulse pressure in CKD and ESRD. Kidney Int. 2012 Aug;82(4):388-400. doi: 10.1038/ki.2012.131. PMID 22534962
- [Background] Georgianos PI, Sarafidis PA, Lasaridis AN. Arterial stiffness: a novel cardiovascular risk factor in kidney disease patients. Curr Vasc Pharmacol. 2015;13(2):229-38. doi: 10.2174/15701611113119990147. PMID 24007427
- [Background] Blacher J, Guerin AP, Pannier B, Marchais SJ, Safar ME, London GM. Impact of aortic stiffness on survival in end-stage renal disease. Circulation. 1999 May 11;99(18):2434-9. doi: 10.1161/01.cir.99.18.2434. PMID 10318666
- [Background] Sipahioglu MH, Kucuk H, Unal A, Kaya MG, Oguz F, Tokgoz B, Oymak O, Utas C. Impact of arterial stiffness on adverse cardiovascular outcomes and mortality in peritoneal dialysis patients. Perit Dial Int. 2012 Jan-Feb;32(1):73-80. doi: 10.3747/pdi.2010.00186. Epub 2011 Mar 31. PMID 21454392
- [Background] Szeto CC, Kwan BC, Chow KM, Leung CB, Law MC, Li PK. Prognostic value of arterial pulse wave velocity in peritoneal dialysis patients. Am J Nephrol. 2012;35(2):127-33. doi: 10.1159/000335580. Epub 2012 Jan 11. PMID 22236995
- [Background] Briet M, Collin C, Karras A, Laurent S, Bozec E, Jacquot C, Stengel B, Houillier P, Froissart M, Boutouyrie P; Nephrotest Study Group. Arterial remodeling associates with CKD progression. J Am Soc Nephrol. 2011 May;22(5):967-74. doi: 10.1681/ASN.2010080863. Epub 2011 Apr 14. PMID 21493771
- [Background] Kimoto E, Shoji T, Shinohara K, Hatsuda S, Mori K, Fukumoto S, Koyama H, Emoto M, Okuno Y, Nishizawa Y. Regional arterial stiffness in patients with type 2 diabetes and chronic kidney disease. J Am Soc Nephrol. 2006 Aug;17(8):2245-52. doi: 10.1681/ASN.2005101038. Epub 2006 Jul 12. PMID 16837632
- [Background] Townsend RR, Wimmer NJ, Chirinos JA, Parsa A, Weir M, Perumal K, Lash JP, Chen J, Steigerwalt SP, Flack J, Go AS, Rafey M, Rahman M, Sheridan A, Gadegbeku CA, Robinson NA, Joffe M. Aortic PWV in chronic kidney disease: a CRIC ancillary study. Am J Hypertens. 2010 Mar;23(3):282-9. doi: 10.1038/ajh.2009.240. Epub 2009 Dec 17. PMID 20019670
- [Background] Guerin AP, Blacher J, Pannier B, Marchais SJ, Safar ME, London GM. Impact of aortic stiffness attenuation on survival of patients in end-stage renal failure. Circulation. 2001 Feb 20;103(7):987-92. doi: 10.1161/01.cir.103.7.987. PMID 11181474
- [Background] Jung JY, Hwang YH, Lee SW, Lee H, Kim DK, Kim S, Oh YG, Yang J, Joo KW, Ahn C, Oh KH. Factors associated with aortic stiffness and its change over time in peritoneal dialysis patients. Nephrol Dial Transplant. 2010 Dec;25(12):4041-8. doi: 10.1093/ndt/gfq293. Epub 2010 May 25. PMID 20501463
- [Background] Utescu MS, Couture V, Mac-Way F, De Serres SA, Marquis K, Lariviere R, Desmeules S, Lebel M, Boutouyrie P, Agharazii M. Determinants of progression of aortic stiffness in hemodialysis patients: a prospective longitudinal study. Hypertension. 2013 Jul;62(1):154-60. doi: 10.1161/HYPERTENSIONAHA.113.01200. Epub 2013 May 6. PMID 23648699
- [Background] Agarwal R. Arterial stiffness and its relationship to clinic and ambulatory blood pressure: a longitudinal study in non-dialysis chronic kidney disease. Nephrol Dial Transplant. 2017 Nov 1;32(11):1850-1856. doi: 10.1093/ndt/gfw281. PMID 27474747
- [Background] Agarwal R, Brim NJ, Mahenthiran J, Andersen MJ, Saha C. Out-of-hemodialysis-unit blood pressure is a superior determinant of left ventricular hypertrophy. Hypertension. 2006 Jan;47(1):62-8. doi: 10.1161/01.HYP.0000196279.29758.f4. Epub 2005 Dec 12. PMID 16344376
- [Background] Agarwal R, Peixoto AJ, Santos SF, Zoccali C. Pre- and postdialysis blood pressures are imprecise estimates of interdialytic ambulatory blood pressure. Clin J Am Soc Nephrol. 2006 May;1(3):389-98. doi: 10.2215/CJN.01891105. Epub 2006 Apr 12. PMID 17699236
- [Background] Georgianos PI, Agarwal R. Epidemiology, diagnosis and management of hypertension among patients on chronic dialysis. Nat Rev Nephrol. 2016 Oct;12(10):636-47. doi: 10.1038/nrneph.2016.129. Epub 2016 Aug 30. PMID 27573731
- [Background] Atas N, Erten Y, Okyay GU, Inal S, Topal S, Onec K, Akyel A, Celik B, Tavil Y, Bali M, Arinsoy T. Left ventricular hypertrophy and blood pressure control in automated and continuous ambulatory peritoneal dialysis patients. Ther Apher Dial. 2014 Jun;18(3):297-304. doi: 10.1111/1744-9987.12104. PMID 24965296
- [Background] Jang JS, Kwon SK, Kim HY. Comparison of Blood Pressure Control and Left Ventricular Hypertrophy in Patients on Continuous Ambulatory Peritoneal Dialysis (CAPD) and Automated Peritoneal Dialysis (APD). Electrolyte Blood Press. 2011 Jun;9(1):16-22. doi: 10.5049/EBP.2011.9.1.16. Epub 2011 Jun 30. PMID 21998602
- [Background] Koc M, Toprak A, Tezcan H, Bihorac A, Akoglu E, Ozener IC. Uncontrolled hypertension due to volume overload contributes to higher left ventricular mass index in CAPD patients. Nephrol Dial Transplant. 2002 Sep;17(9):1661-6. doi: 10.1093/ndt/17.9.1661. PMID 12198220
- [Background] O'Shaughnessy MM, Durcan M, Kinsella SM, Griffin MD, Reddan DN, Lappin DW. Blood pressure measurement in peritoneal dialysis: which method is best? Perit Dial Int. 2013 Sep-Oct;33(5):544-51. doi: 10.3747/pdi.2012.00027. Epub 2013 Apr 1. PMID 23547279
- [Background] Wang MC, Tseng CC, Tsai WC, Huang JJ. Blood pressure and left ventricular hypertrophy in patients on different peritoneal dialysis regimens. Perit Dial Int. 2001 Jan-Feb;21(1):36-42. PMID 11280494
- [Background] Nakahigashi M, Tsukaguchi H, Morimoto S, Nakano C, Ueda H, Someya K, Kusabe M, Kikuchi S, Imada T, Shiojima I. Determinants of the Change in Arterial Stiffness in Peritoneal Dialysis Patients. Int Heart J. 2017 Dec 12;58(6):915-925. doi: 10.1536/ihj.16-624. Epub 2017 Nov 17. PMID 29151492
- [Background] London GM, Pannier B. Arterial functions: how to interpret the complex physiology. Nephrol Dial Transplant. 2010 Dec;25(12):3815-23. doi: 10.1093/ndt/gfq614. Epub 2010 Oct 14. PMID 20947536
- [Background] Protogerou AD, Papaioannou TG, Blacher J, Papamichael CM, Lekakis JP, Safar ME. Central blood pressures: do we need them in the management of cardiovascular disease? Is it a feasible therapeutic target? J Hypertens. 2007 Feb;25(2):265-72. doi: 10.1097/HJH.0b013e3280114f23. PMID 17211229
- [Background] Vlachopoulos C, Aznaouridis K, O'Rourke MF, Safar ME, Baou K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with central haemodynamics: a systematic review and meta-analysis. Eur Heart J. 2010 Aug;31(15):1865-71. doi: 10.1093/eurheartj/ehq024. Epub 2010 Mar 2. PMID 20197424
- [Background] Asmar RG, London GM, O'Rourke ME, Safar ME; REASON Project Coordinators and Investigators. Improvement in blood pressure, arterial stiffness and wave reflections with a very-low-dose perindopril/indapamide combination in hypertensive patient: a comparison with atenolol. Hypertension. 2001 Oct;38(4):922-6. doi: 10.1161/hy1001.095774. PMID 11641310
- [Background] Williams B, Lacy PS, Thom SM, Cruickshank K, Stanton A, Collier D, Hughes AD, Thurston H, O'Rourke M; CAFE Investigators; Anglo-Scandinavian Cardiac Outcomes Trial Investigators; CAFE Steering Committee and Writing Committee. Differential impact of blood pressure-lowering drugs on central aortic pressure and clinical outcomes: principal results of the Conduit Artery Function Evaluation (CAFE) study. Circulation. 2006 Mar 7;113(9):1213-25. doi: 10.1161/CIRCULATIONAHA.105.595496. Epub 2006 Feb 13. PMID 16476843
- [Background] Protogerou AD, Argyris A, Nasothimiou E, Vrachatis D, Papaioannou TG, Tzamouranis D, Blacher J, Safar ME, Sfikakis P, Stergiou GS. Feasibility and reproducibility of noninvasive 24-h ambulatory aortic blood pressure monitoring with a brachial cuff-based oscillometric device. Am J Hypertens. 2012 Aug;25(8):876-82. doi: 10.1038/ajh.2012.63. Epub 2012 Jun 7. PMID 22673021
- [Background] Wassertheurer S, Kropf J, Weber T, van der Giet M, Baulmann J, Ammer M, Hametner B, Mayer CC, Eber B, Magometschnigg D. A new oscillometric method for pulse wave analysis: comparison with a common tonometric method. J Hum Hypertens. 2010 Aug;24(8):498-504. doi: 10.1038/jhh.2010.27. Epub 2010 Mar 18. PMID 20237499
- [Background] Weber T, Wassertheurer S, Rammer M, Maurer E, Hametner B, Mayer CC, Kropf J, Eber B. Validation of a brachial cuff-based method for estimating central systolic blood pressure. Hypertension. 2011 Nov;58(5):825-32. doi: 10.1161/HYPERTENSIONAHA.111.176313. Epub 2011 Sep 12. PMID 21911710
- [Background] Sarafidis PA, Georgianos PI, Karpetas A, Bikos A, Korelidou L, Tersi M, Divanis D, Tzanis G, Mavromatidis K, Liakopoulos V, Zebekakis PE, Lasaridis A, Protogerou AD. Evaluation of a novel brachial cuff-based oscillometric method for estimating central systolic pressure in hemodialysis patients. Am J Nephrol. 2014;40(3):242-50. doi: 10.1159/000367791. Epub 2014 Oct 11. PMID 25322847
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] Parati G, Stergiou GS, Asmar R, Bilo G, de Leeuw P, Imai Y, Kario K, Lurbe E, Manolis A, Mengden T, O'Brien E, Ohkubo T, Padfield P, Palatini P, Pickering T, Redon J, Revera M, Ruilope LM, Shennan A, Staessen JA, Tisler A, Waeber B, Zanchetti A, Mancia G; ESH Working Group on Blood Pressure Monitoring. European Society of Hypertension guidelines for blood pressure monitoring at home: a summary report of the Second International Consensus Conference on Home Blood Pressure Monitoring. J Hypertens. 2008 Aug;26(8):1505-26. doi: 10.1097/HJH.0b013e328308da66. PMID 18622223
- [Background] London GM, Pannier B, Guerin AP, Blacher J, Marchais SJ, Darne B, Metivier F, Adda H, Safar ME. Alterations of left ventricular hypertrophy in and survival of patients receiving hemodialysis: follow-up of an interventional study. J Am Soc Nephrol. 2001 Dec;12(12):2759-2767. doi: 10.1681/ASN.V12122759. PMID 11729246
- [Derived] Vareta G, Georgianos PI, Vaios V, Sgouropoulou V, Georgianou EI, Leivaditis K, Mavromatidis K, Dounousi E, Papagianni A, Balaskas EV, Zebekakis PE, Liakopoulos V. Prevalence of Apparent Treatment-Resistant Hypertension in ESKD Patients Receiving Peritoneal Dialysis. Am J Hypertens. 2022 Nov 2;35(11):918-922. doi: 10.1093/ajh/hpac086. PMID 35882382